CLINICAL TRIAL: NCT00600639
Title: Non-Invasive Mechanical Ventilation in Elderly Patients Affected by Acute Hypercapnic Respiratory Failure:A Randomized Control Study vs Standard Medical Therapy A Multicentric Randomized Controlled Trial
Brief Title: Non-Invasive Mechanical Ventilation in Elderly Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Collaborators: Villa Gaiato, Modena (Unknown); Ospedale Regionale di Locarno (Other)
Responsible Party: Fondazione S.Maugeri
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FSM2004-78; 2004-78
Record Dates: First submitted 2008-01-14; First posted 2008-01-25 (Estimated); Last update posted 2012-07-17 (Estimated); Status verified 2008-01

CONDITIONS: Acute Respiratory Failure
Keywords: old patients; NIV; Intubation; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Prednisolone; Anti-Bacterial Agents; Health Services Needs and Demand

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): non-invasive ventilation with BiPAP Vision or another ICU ventilator with NIV option
  Interventions: Device: Non-invasive mechanical ventilation using a BiPAP Vision or any other ICU ventilators with NIV option; Drug: standard medical therapy plus oxygen that includes salbutamol, prednisolone and antibiotics as needed
- 2 (Active Comparator): standard therapy + oxygen
  Interventions: Drug: standard medical therapy that includes salbutamol, prednisolone and antibiotics as needed

INTERVENTIONS:
Device: Non-invasive mechanical ventilation using a BiPAP Vision or any other ICU ventilators with NIV option — A mode of ventilation that does not require the insertion of the endotracheal tube, since the support is delivered throgh a full face or nasal mask
  Other Names: BiPAP Vision or any other ICU ventilators with NIV option
  Arms: 1
Drug: standard medical therapy plus oxygen that includes salbutamol, prednisolone and antibiotics as needed — Standard medical therapy includes drugs like beta2-agonists, steroids, anthicolinergic agents- antibuiotics as needed
  Arms: 1
Drug: standard medical therapy that includes salbutamol, prednisolone and antibiotics as needed — oxygen plus medical therapy for ARF
  Arms: 2

SUMMARY:
The efficacy of NIMV to treat HARF has been widely demonstrated. However, in most of the studies performed in ICUs and in another facilities the mean age of the patients is usually less than 70 years.

A multicentric, randomized-controlled trial conduced in a group of "ELDERLY" patients with the mean age higher than 76 years, to compare the use of NIMV with Standard Medical Treatment (SMT) in the treatment of an episode of Acute Hypercapnic Respiratory Failure.

DETAILED DESCRIPTION:
Non-invasive mechanical ventilation (NIMV) has been successfully used in Hypercapnic Acute Respiratory Failure (HARF) since endotracheal intubation (ETI) and invasive ventilation are associated to high morbidity and mortality rate.

because of the lack of beds in most Intensive Care Units (ICUs) and the high mortality and cost associated with the increased of age, the "Elderly" patients affected by ARF due to chronic diseases are not always considered for ETI.

The efficacy of NIMV to treat HARF has been widely demonstrated. However, in most of the studies performed in ICUs and in another facilities the mean age of the patients is usually less than 70 years (see tab1).

Authors MEAN AGE

(yrs) TYPE of STUDY

Bott <80 COPD NIV vs Medical Therapy

Brochard71±9 COPD NIV vs Medical Therapy

Kramer 66±7 COPD NIV vs Medical Therapy

Andeev 63±4 COPD NIV vs Medical Therapy

Barbe 70±2 COPD NIV vs Medical Therapy

Bardi 68±8 COPD NIV vs Medical Therapy

Plant 69±8 COPD NIV vs Medical Therapy

Thys 71±8 COPD NIV vs sham NIV

Nava 68±8 COPD NIV in weaning

Girault 63±14 NIV in weaning

Ferrer 70±7 NIV in weaning

Hill 71±3 COPD PAV vs PSV

Confalonieri 66±14 PNEUMONIA NIV vs Medical Therapy

Martin 64±17 Miscellaneous NIV vs Medical Therapy

Conti 72±7 COPD NIV vs EI

A multicentric, randomized-controlled trial conducted in a group of "ELDERLY" patients with the mean age higher than 76 years, to compare the use of NIMV with Standard Medical Treatment (SMT) in the treatment of an episode of Acute Hypercapnic Respiratory Failure.

ELIGIBILITY:
Inclusion Criteria:

* Age higher 75 years old
* Hypercapnic acute respiratory failure (PaCO2 greater 50 mmHg and pH lower than 7.35)
* Respiratory rate (RR) higher 25 bpm after 12 hours of standard medical therapy.

Exclusion Criteria:

* Respiratory failure due to pulmonary oedema
* Kelly's score equal or higher than 4
* Cardio-respiratory arrest
* Systolic arterial blood pressure greater than 90 mmHg or severe arrhythmia
* Recent facial, oesophageal and gastric surgery

Min Age: 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 82 (Actual)
Dates: Start 2004-01; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Meet the criteria for INTUBATION: pH < 7.2 or pH < 7.25 in two consecutive occasions or worsening pH during NIV or rapid increase of 20mmHg of PaCO2 from baseline or PaO2< 50mmHg with FiO2 40% or Kelly score > 4 Mortality rate | 3 months

SECONDARY OUTCOMES:
Arterial Blood Gasses improvement Clinical improvement (decrease of respiratory rate and dyspnoea value) Length of Hospital stay | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Nava, Principal Investigator — Fondazione Salvatore Maugeri
Locations (1):
- Istituto Scientifico di Pavia Fondazione Salvatore Maugeri, Pavia, Pavia, Italy